CLINICAL TRIAL: NCT05102474
Title: Dermatologic Research Evaluation and Monitoring of Sleep in Moderate-to-Severe Psoriasis
Acronym: DREAMS-PSO
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis Pharmaceuticals (Industry); National Psoriasis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: DREAMS-PSO
Record Dates: First submitted 2021-10-18; First posted 2021-11-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate to Severe Psoriasis: Moderate to severe psoriasis will be defined as affected body surface area (BSA) ≥3%.
  Interventions: Other: Polysomnography (PSG)
- Healthy Controls: Healthy controls will be age and sex matched subjects with no prior or current history of psoriasis.
  Interventions: Other: Polysomnography (PSG)

INTERVENTIONS:
Other: Polysomnography (PSG) — PSG is the gold standard for objectively measuring sleep in the laboratory setting. The procedure consists of electrodes measuring brain activity (electroencephalography, EEG), eye movements (electrooculography, EOG), muscle activity (electromyography, EMG), respiratory events, snoring activity, blood oxygen saturation, and body position. Video surveillance during the sleep study can also monitor for itching events that occur during the night.

SUMMARY:
Getting enough sleep is important for maximizing health and well-being. When it comes to health, sleep is as vital as regular exercise and eating a balanced diet. Not getting enough sleep can lead to health problems like heart attacks, diabetes, and even cancer. Since individuals with psoriasis have these same health problems, getting better sleep may help to keep them happier and healthier. This study will look at how individuals with psoriasis sleep and if their sleep is different than indivuduals without psoriasis.

DETAILED DESCRIPTION:
A growing body of literature has revealed that individuals with psoriasis are more likely to report sleep disturbance when compared to the general population. The cross-sectional study presented here will allow the investigators to objectively and rigorously measure sleep architecture in psoriasis patients and compare it to healthy controls, If sleep dysfunction is confirmed in this population, then clinical interventions such as screening for sleep disturbance or promoting sleep hygiene could lead to meaningful improvements in patients' health, longevity, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of moderate to severe plaque type psoriasis confirmed by the principal investigator. Moderate to severe psoriasis will be defined as affected BSA ≥3%. Healthy controls will be age and sex matched (see below) subjects with no prior or current history of psoriasis.
2. Are at least 18 years of age
3. Psoriasis has been stable over the last 3 months
4. Psoriasis is either untreated or treated only with topicals at the current time (see exclusion criteria for washout times)
5. Subjectively reported poor sleep quality using the Pittsburg Sleep Quality Index (PSQI) (defined as a global score >5)
6. Fluent in English
7. Demonstrate understanding of the study and willingness to participate as evidenced by voluntary informed consent

Exclusion Criteria:

1. Patients with guttate, erythrodermic, or pustular psoriasis subtypes
2. Having a previous diagnosis of obstructive sleep apnea (OSA) or another medically defined sleep disorder or fall into the intermediate or high-risk groups for having OSA as calculated by the STOP-BANG questionnaire
3. Subjects who have used the following treatments for psoriasis: phototherapy (UVB) in the last 2 weeks, photochemotherapy (PUVA) in the last 4 weeks, oral systemic treatments in the last 4 weeks, biologic immunomodulating agents in the last 12 weeks, or have had exposure to any other investigational drug/device within 30 days prior to study entry
4. Subjects who have used any over the counter or prescription sleep aids within five half-lives of the agent in question.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 24 patients (12 moderate-to-severe psoriasis and 12 healthy controls, age and sex matched) will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency | Average over 3 consecutive nights of sleep
  Sleep efficiency is defined as the percentage of time spent asleep while in bed.

SECONDARY OUTCOMES:
Total sleep time | Average over 3 consecutive nights of sleep
  Total sleep time is the total amount of sleep time recorded during the total recording time (each night)
Sleep onset latency | Average over 3 consecutive nights of sleep
  Sleep onset latency is defines as the duration of time from turning off the light to falling asleep.
Wake after sleep onset | Average over 3 consecutive nights of sleep
  Wake after sleep onset is defined as the time between when they first fall asleep to when they become fully awake.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Bhutani, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psorisis Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No